CLINICAL TRIAL: NCT02098915
Title: The Use of Metoclopramide vs. Placebo in Infants With Gastroschisis. A Pilot Double Blind Randomized Controlled Trial
Brief Title: Metoclopramide Pilot Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision to prematurely close the trial was made because of poor recruitment.
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Jacob Langer, Jacob C Langer, MD, FRCSC, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000038585; 169334 (Other: Health Canada)
Record Dates: First submitted 2014-03-21; First posted 2014-03-28 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Gastroschisis
Keywords: gastroschisis; intestinal motility; prokinetic agents; intravenous metoclopramide; time to full enteral feeding
MeSH Terms: conditions — Gastroschisis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intravenous metoclopramide (Experimental): the experimental arm will receive intravenous metoclopramide
  Interventions: Drug: intravenous metoclopramide
- control arm (Placebo Comparator): the control arm will receive placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: intravenous metoclopramide — the experimental arm will receive intravenous metoclopramide dosed according to the current Sick Kids guidelines based upon weight and age
  Arms: intravenous metoclopramide
Other: Placebo — equivalent volume to intravenous metoclopramide (dosed according to the current Sick Kids guidelines based upon weight and age ) of sterile sodium chloride 0.9% injection as a placebo
  Arms: control arm

SUMMARY:
Infants with gastroschisis typically have poor intestinal motility for the first weeks to months after birth. Prokinetic agents are often used in these infants to improve intestinal motility in an attempt to quicken the attainment of enteric feeds. However, the evidence to support this practice remains weak. Investigators hypothesize that a prokinetic agent given intravenously (infused into a vein) may be effective in improving gut motility in children with gastroschisis.

DETAILED DESCRIPTION:
The research question will be addressed in a pilot randomized double-blind placebo controlled clinical trial evaluating the efficacy of metoclopramide.Investigators will recruit 30 neonates (15 per arm) diagnosed with gastroschisis. There will be two arms to the trial: the experimental arm will receive intravenous metoclopramide and the control arm will receive placebo. Patients will receive prokinetic agent therapy, dosed according to weight, or placebo. Each subject will receive the intervention for 28 days or until achievement of full enteral feeding, whichever comes first. Primary outcome: Days to achieve full enteral feeding when all intake (at least 150 ml/kg/day for 72 hours) is given as breast milk or formula by gavage or by mouth. Secondary outcomes: 1. Duration (days) until initiation of enteral feeds. 2. Duration (days) on parenteral nutrition. 3. Weight gain, measured by grams per day per week during therapy. 4. Occurrence of adverse effects associated with the use of metoclopramide. 5. Rate of catheter-related sepsis episodes (line positive blood cultures necessitating antibiotic treatment or catheter removal). 6. Incidence of necrotizing enterocolitis (NEC) based on clinical criteria and presence of pneumatosis intestinalis on an abdominal X-ray. 7. Duration of hospitalization (number of days from admission until final hospital discharge).

Subjects can be withdrawn from the study if meet one of the following criteria:

* Subject develops extrapyramidal symptoms
* Subject has not established full enteral feeding by the end of day 28 of therapy
* Withdrawal of informed consent or refusal of further study participation by parent/legal guardian
* Serious adverse event which, in the opinion of the investigator, indicates that continued participation in the study is not in the best interest of the subject
* Any clinical adverse event, laboratory abnormality or intercurrent illness which, in the opinion of the investigator, indicates that continued participation in the study is not in the best interest of the subject
* Unpredictable discontinuation of metoclopramide drug supply

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of uncomplicated neonatal gastroschisis treated by primary fascial closure or delayed closure using a pre-formed silo (fascial closure or plastic closure)
2. Expectation of the treating physician that the patient will require intravenous therapy for at least 7 days post-enrolment

Exclusion Criteria:

1. Presence of other significant congenital malformation (ie life-threatening, requiring surgical intervention, or having an effect on intestinal motility)
2. Presence of intestinal atresia, intestinal necrosis or intestinal perforation (ie complicated gastroschisis)
3. Gestational age <32 weeks
4. Birth weight < 1500 gm
5. Received an investigational product within the past 30 days

Min Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Days to achieve full enteral feeding | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 4 weeks. Days to achieve full enteral feeding will be recorded when all intake (at least 150 ml/kg/day for 72 hours) is given as breast milk or formula by gavage or by mouth

SECONDARY OUTCOMES:
Duration until initiation of enteral feeds | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 4 weeks. Duration (days) until initiation of enteral feeds will be recorded
Duration on parenteral nutrition | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 4 weeks. Duration (days) on parenteral nutrition will be recorded
Weight gain | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 4 weeks. Weight gain, measured by grams per day per week during therapy will be recorded
Occurrence of adverse effects | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 4 weeks. Occurrence of adverse effects associated with the use of metoclopramide will be recorded.
Rate of catheter-related sepsis episodes | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 4 weeks. Rate of catheter-related sepsis episodes during intravenous treatment (line positive blood cultures necessitating antibiotic treatment or catheter removal) will be recorded.
Incidence of necrotizing enterocolitis (NEC) | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 4 weeks. Incidence of necrotizing enterocolitis (NEC) during the therapy based on clinical criteria and presence of pneumatosis intestinalis on an abdominal X-ray will be recorded.
Duration of hospitalization | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Duration of hospitalization (number of days from admission until final hospital discharge) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob C Langer, MD, Principal Investigator — University of Toronto
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada